CLINICAL TRIAL: NCT02218827
Title: Evaluation of Steroidal Treatment For Dry Eye Disease
Brief Title: Topical Steroid Treatment For Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, shay ofir, Medical Doctir, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: dry eye01
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Dry Eye
Keywords: Dry Eye; Inflammatory reaction; steroids
MeSH Terms: conditions — Dry Eye Syndromes; Inflammation | interventions — Loteprednol Etabonate; Fluorometholone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dry eye patients (Experimental): Loteprednol Etabonate (FML) topical treatment 1 drop 4 times daily for 1 month then Loteprednol Etabonate (FML) 1 drop 2 times daily for 1 month
  Interventions: Drug: Loteprednol Etabonate (FML)

INTERVENTIONS:
Drug: Loteprednol Etabonate (FML) — a steroid topical treatment used for moderate dry eye symptoms. this drug causes less increase in intra ocular pressure

SUMMARY:
Many patients refer to an oculoplastic or corneal clinic examination due to dry eye symptoms. epidemiologic studies estimate that as many as 15% of the population over 60 years suffer from dry eye. the disease can be treated both topically through several drugs or through mechanical closure of the lacrimal drainage system. in the past decade a few studies demonstrated the efficacy of anti inflammatory treatment on dry eye disease due to the inflammatory process that occurs in it. this treatment rises goblet cell counts but in the meantime elevates the intra ocular pressure and elevates the risk for infections. steroids that cause a lower increase in intraocular pressure have not been thoroughly evaluated in dry eye disease. we with to subjectively and objectively evaluate an FDA approved topical steroidal drug in the treatment of dry eye.

DETAILED DESCRIPTION:
30 patients 21 year or older, from both sexes with no previous eyelid or corneal surgeries, refered to our outpatient clinics will be recruited and evaluated.

the initial examination will include schirmer1 test, Tear break up time test, a full ophthalmologic evaluation and a dry eye questionaire.

after signing a concent form patient will be treated with Loteprednol Etabonate four times a ady for a month, then a second examination will take place. after that and according to necessity patients will be treated with Loteprednol Etabonate two times daily for another month and return for a follow up examination. intraocular pressure will be evaluated in each follow up visit as well as dry eye symptoms, schirmer 1 test and tear break up time test.

ELIGIBILITY:
Inclusion Criteria:

* referral for ophthalmic examination due to dry eye symptoms
* ability to sign a concent form

Exclusion Criteria:

* former corneal, eyelid or lacrimal gland operations
* former orbital chemotherapy or irradiation treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
clinical improvement in dry eye measurements | two months
  tear break up time and schirmer 1 test will evaluate improvement in dry eye under medical treatment

SECONDARY OUTCOMES:
symptomatic improvement | two months
  dry eye questionaire will be evaluated on each follow up

CONTACTS AND LOCATIONS:
Overall Officials: Shay Ofir, Dr, Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - Meir Medical center, Kfar Saba, Israel
  - Sheba Medical Center, Ramat Gan